CLINICAL TRIAL: NCT03505060
Title: A Phase 1b Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of the IHV01 Protein Vaccine Primed and Co-administered With HIV DNA CON-S Env Vaccine in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of the IHV01 Protein Vaccine Primed and Co-Administered With HIV DNA CON-S Env Vaccine in Healthy, HIV-1-Uninfected Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: One of the study products is no longer available for clinical trial use.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 125; 30015 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: DNA CON-S env + IHV01 (Experimental): Participants will receive 4 mg of DNA CON-S env at Months 0 and 1. They will receive 4 mg of DNA CON-S env and 150 mcg of IHV01 at Months 3 and 6.
  Interventions: Biological: DNA CON-S env; Biological: IHV01
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo at Months 0, 1, 3, and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DNA CON-S env — Administered by intramuscular injection in the deltoid.
  Arms: Group 1: DNA CON-S env + IHV01
Biological: IHV01 — Administered by intramuscular injection in the deltoid.
  Arms: Group 1: DNA CON-S env + IHV01
Biological: Placebo — Sodium Chloride for Injection, USP 0.9%; administered by intramuscular injection in the deltoid.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the IHV01 protein vaccine primed and co-administered with HIV DNA CON-S env vaccine in healthy, HIV-1-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of the IHV01 protein vaccine primed and co-administered with HIV DNA CON-S env vaccine in healthy, HIV-1-uninfected adults.

Participants will be randomly assigned to two groups. Participants in Group 1 will receive 4 mg of DNA CON-S env at Months 0 and 1. They will receive 4 mg of DNA CON-S env and 150 mcg of IHV01 at Months 3 and 6. Participants in Group 2 will receive placebo at Months 0, 1, 3, and 6.

Study visits will occur at Day 0 (study entry), Week 2, and Months 1, 1.5, 3, 3.5, 6, 6 + 1 week, 6.5, and 12. Visits may include physical examinations, medical history, injection of study product, blood and urine collection, pregnancy testing, HIV testing, risk reduction counseling, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last required clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit. Low risk guidelines are found on the protocol web page under Study Materials on the HVTN Members' site (https://members.hvtn.org/protocols/hvtn125).

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal and creatinine less than or equal to institutional upper limits of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

Normal urine:

* Negative urine glucose, and
* Negative or trace urine protein, and
* Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until three months after the last study injection. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 125 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 125 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 125 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 125 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made by the HVTN 125 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 125 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 125 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than or equal to 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment)
* Serious adverse reactions to vaccines or to vaccine components such as mannitol and aluminum hydroxide, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination (for mAb see related criterion above)
* Autoimmune disease (Not exclusionary: mild, well-controlled psoriasis)
* Immunodeficiency

Clinically significant medical conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-11-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of local and systemic reactogenicity signs and symptoms | Measured through 1 week after the last vaccination (Month 6 + 1 week)
  Systemic symptoms may include increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, and nausea. Local symptoms include pain and/or tenderness at the injection site. All reactogenicity symptoms are graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, except as noted in the protocol.
Distribution of values of laboratory measures of safety | Measured through Month 12
  Based on laboratory evaluations (graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017)
Frequency of adverse events (AEs) | Measured through Month 12
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Frequency of serious adverse events (SAEs) | Measured through Month 12
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Change in Env-specific IgG binding response rate | Measured through Month 6.5
  Measured by binding antibody assays

SECONDARY OUTCOMES:
Change in magnitude of Env-specific IgG binding antibodies | Measured through Month 6.5
  Measured by binding antibody assays
Change in response rate of antibody-dependent cellular cytotoxicity (ADCC)-mediating antibody responses | Measured through Month 6.5
  Assessed using serum samples taken at the primary immunogenicity time point
Change in response rate of antibody-dependent cellular phagocytosis (ADCP)-mediating antibody responses | Measured through Month 6.5
  Measured using serum/plasma samples taken at baseline and primary immunogenicity timepoints
Change in response rate of Env-specific CD4+ and CD8+ T-cell responses | Measured at Month 6.5
  Measured by intracellular cytokine staining (ICS)
Change in magnitude of pTfh response | Measured through 1 week after the last vaccination (Month 6 + 1 week)
  Measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchbinder, Study Chair — San Francisco Department of Public Health; Sonya Heath, Study Chair — University of Alabama at Birmingham
Locations (1):
- Bridge HIV CRS, San Francisco, California, United States